CLINICAL TRIAL: NCT04979455
Title: Prospective Investigation of Risk Factors for Exertional Heat Illness
Brief Title: Risk Factors for Exertional Heat Illness
Status: Active, not recruiting | Type: Observational
Sponsor: Liverpool John Moores University (Other)
Collaborators: Institute of Naval Medicine (UK) (Unknown); CTCRM Lympstone (UK) (Unknown); University of Portsmouth (UK) (Unknown); Public Health Wales (Other Government); Bangor University (UK) (Unknown); Headquarters Army Recruiting and Initial Training Command (UK) (Unknown); Defence Science and Technology (UK) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2029/MODREC/21
Record Dates: First submitted 2021-05-28; First posted 2021-07-28 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-10

CONDITIONS: Exertional Heat Illness
MeSH Terms: conditions — Heat Stress Disorders | interventions — Surveys and Questionnaires; Urine Specimen Collection; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva sample, stool sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Exertional heat illness: Participants who experience an atypical elevation in thermal strain or an EHI undergoing strenuous physical exercise.
  Interventions: Other: Core temperature monitoring; Behavioral: Questionnaires; Other: Heart rate monitoring; Other: Urine collection; Other: Sleep monitoring; Other: Blood collection; Other: Saliva collection; Other: Throat swab collection; Other: Stool collection
- Control: Participants who do not experience an atypical elevation in thermal strain or an EHI undergoing strenuous physical exercise.
  Interventions: Other: Core temperature monitoring; Behavioral: Questionnaires; Other: Heart rate monitoring; Other: Urine collection; Other: Sleep monitoring; Other: Blood collection; Other: Saliva collection; Other: Throat swab collection; Other: Stool collection

INTERVENTIONS:
Other: Core temperature monitoring — Core temperature will be monitored on the day of exercise
Behavioral: Questionnaires — Questionnaires will be completed at baseline and on the day of exercise
Other: Heart rate monitoring — Heart rate will be monitored on the day of exercise
Other: Urine collection — Urine samples will be collected at baseline and on the day of exercise
Other: Sleep monitoring — Sleep will be monitored at baseline and on the day of exercise
Other: Blood collection — Blood samples will be completed at baseline
Other: Saliva collection — Saliva samples will be collected at baseline and on the day of exercise
Other: Throat swab collection — Throat swab samples will be collected at baseline and on the day of exercise
Other: Stool collection — Stool samples will be collected at baseline and on the day of exercise

SUMMARY:
The arduous nature of military training and operations require personnel to encounter high heat load, e.g., during intense physical exertion, particularly in the heat. These conditions reduce operational effectiveness and expose personnel to a risk of incapacitation and death from exertional heat illness (EHI).

The aim of this study is to examine traditional and novel risk factors that may increase thermal strain and EHI likelihood in military recruits undergoing strenuous physical exercise.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 17-35 years enrolled in military training

Exclusion Criteria:

* Self-report as pregnant

Ages: 17 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants who experience and participants who do not experience an atypical elevation in thermal strain or an EHI undergoing strenuous physical exercise.
Sampling Method: Non-Probability Sample
Enrollment: 783 (Estimated)
Dates: Start 2021-06-11 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Body mass index in EHI and control group | Baseline
Fitness in EHI and control group - participants ranked by time to complete fitness test | Baseline
Core temperature in EHI and control group | 1 Day
Heart rate in EHI and control group | 2 Hours
Urine osmolality in EHI and control group | Baseline
Sleep quality and quantity, measured by Pittsburgh Sleep Quality Index, in EHI and control group | Throughout study - up to 1 week
  0-21 Scale. Higher score indicates worse outcome
Sleep quality, measured by actigraphy, between EHI and control group | Throughout study - up to 1 week
Sleep quantity, measured by actigraphy, between EHI and control group | Throughout study - up to 1 week
Circulating Interleukin 6 in EHI and control group | Baseline
Circulating C-Reactive Protein in EHI and control group | Baseline
Circulating Creatine kinase in EHI and control group | Baseline
Circulating Aspartate Aminotransferase in EHI and control group | Baseline
Circulating Alanine Aminotransferase in EHI and control group | Baseline
Circulating Claudin 3 in EHI and control group | Baseline
Circulating Zonulin in EHI and control group | Baseline
Circulating Lipopolysaccharide binding protein in EHI and control group | Baseline
Circulating immunoglobulin E in EHI and control group | Baseline
Salivary cortisol in EHI and control group | Throughout study - up to 1 week
Detection of infectious pathogens in EHI and control groups | Throughout study - up to 1 week
Respiratory illness symptomology, measured by Jackson common cold questionnaire, in EHI and control group | Throughout study - up to 1 week
  0-24 Scale. Higher score indicates worse outcome
Gastrointestinal illness symptomology, measured by gastrointestinal symptoms questionnaire, in EHI and control group | Throughout study - up to 1 week
  0-10 Scale per symptom. Higher score indicates worse outcome
Abundance and diversity of gastrointestinal microbiota in EHI and control group | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Commando Training Centre Royal Marine, Lympstone, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No